CLINICAL TRIAL: NCT06121817
Title: Thermogenic Effect and Metabolic Responses of Durian
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-052
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Effects of; Food; Thermogenesis; Blood Pressure; Heart Rate
Keywords: Thermic Effect of Food; Blood Glucose; Lipid test; Blood Pressure; Heart Rate; exotic fruits

STUDY DESIGN:
Intervention Model Description: All subjects will have both durian and banana interventions, with a wash-out period of at least 5 days between interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durian (Experimental): 250 g of durian aril (isocaloric)
  Interventions: Other: Food/meal intervention
- Banana (Other): 417.6 g of banana (isocaloric)
  Interventions: Other: Food/meal intervention

INTERVENTIONS:
Other: Food/meal intervention — 2 types of exotic fruits, durian and banana, are the study test meals. Both isocaloric test meals are performed at breakfast. All subjects are required to consume the entire meal within 10 minutes.

SUMMARY:
The primary aim of this study is to determine the effectiveness of durian on thermic effect of food (TEF), blood pressure, heart rate and postprandial glucose and lipid levels in young healthy men and women, compared to the ingestion of isocaloric banana.

DETAILED DESCRIPTION:
Visit 1: Consenting and screening for study criteria. Visit 1 consists of consenting and screening session. Potential subjects will arrive at CNRC at 8h30 after 10-hour overnight fast (at least), only allowed access to water. A copy of written participant information sheet and informed consent form (ICF) will be given for them to read through carefully with needed time, and they may question for unclarity. Upon satisfaction, subjects must sign the ICF prior to the study procedures. After the consent, subjects will be screened for their eligibility with health screening questionnaire, and undergo anthropometric measurements (i.e. weight, height, waist circumference, and hip circumference). BMI will be calculated using formular weight divided by meter square (kg/m2). Blood pressure and heart rate readings will be taken. Body composition will be assessed using bioimpedance (BIA). Female subjects will be required to perform a β-HCG test using a urinary pregnancy test kit. Fasting glucose test will be performed through finger prick.

Visit 2 and 3: Intervention study (durian or banana will be assigned randomly) Visit 2 and visit 3 correspond to test session. Female subjects will be tested in the follicular phase of the menstrual cycle (the last menstrual cycle will be noted during screening and regular follow-up for the update). On each test day, subjects will arrive at CNRC at 8h30 after 10-hour overnight fast (at least), only water is allowed. They will undergo anthropometric measurements, and then instructed to lay comfortably on a bed in a suite (room temperature 22-24°C) for 45-minute of resting metabolic rate (RMR) measurement. Blood pressure, heart rate, fasting blood glucose, and fasting lipid will be performed before the meal test. At 9h30, subjects will be served 250g of durian or 417.6g of banana in a plate with 200 mL of water, and requested to consume the entire test meal within 10 min. Thermic effect of test meal will be performed after ingestion for 3 hours. Blood glucose fluctuation will be measured at 15 min, 30 min, 60 min, 90 min, 120 min, 180 min, and lipid fluctuation will be measured at 60 min, 120 min, and 180 min by finger prick. Blood pressure and heart rate readings will be taken at 30 min, 60 min, 120 min, 180 min.

ELIGIBILITY:
Inclusion Criteria:

* BMI with the range of 18-25 kg/m2
* Aged between 21 and 40 year-old
* Chinese origin
* Non-diabetic, fasting blood glucose ≤ 5.6 mmol/L
* Blood pressure below 140/90 mmHg
* Pass the general health screening questionnaire
* Have a stable bodyweight (<5%) over the past 6 months
* Have no medical history
* Have ability to provide informed consent

Exclusion Criteria:

* Subjects who are smoker or currently on nicotine therapy
* Subjects who regularly consume alcohol (>1 unit per day)
* Subjects who are currently receiving therapy (e.g. insulin) or any medication/treatment (including supplements) that may affect glucose and lipid metabolism, energy metabolism or body composition.
* Subjects who are currently on steroids, protease inhibitors, or antipsychotic therapies
* Subjects who recently had a major medical or surgical event or will have one during the study period
* Subjects who have symptomatic Irritable Bowel Syndrome
* Subjects who have glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Subjects who have active Tuberculosis (TB) or currently receiving treatment for TB
* Subjects who have chronic infection or is known to suffer from or has previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Subjects who participated in drug trial within 3 months before the start of the study
* Subjects who have allergy or intolerant to durian or/and banana
* Subjects who are unwilling to consume durian or banana
* Subjects who are hemophobia, trypanophobia, or claustrophobia
* Subjects (females) who are pregnant (pregnancy test will be performed), lactating, or planning to become pregnant during the study period
* Subjects who do not have adequate fluency in the English language
* Subjects who are unable to understand the study procedures and to sign forms providing written informed consent to participate in the study
* Subjects who are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female subjects will be tested in the follicular phase of the menstrual cycle (the last menstrual cycle will be noted during screening and regular follow-up).
Enrollment: 16 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Thermic effect of food | 3 hours
  Measured using the Indirect calorimetry (canopy hood)
Blood Pressure | 5 timepoints at 0 minute, 30 minutes, 60 minutes, 120 minutes, and 180 minutes
  Measured using an automated instrument (Omron HEM-907)
Heart Rate | 5 timepoints at 0 minute, 30 minutes, 60 minutes, 120 minutes, and 180 minutes
  Measured using an automated instrument (Omron HEM-907)
Postprandial blood glucose levels | 7 timepoints at 0 minute, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, and 180 minutes
  Glucose levels will be measured using a portable glucose analyzer (Hemocue glucose 201 RT).
Postprandial lipid levels | 4 timepoints at 0 minute, 60 minutes, 120 minutes, and 180 minutes
  Triglycerides, Cholesterol, LDL, HDL measured using the Cobas b101 system

CONTACTS AND LOCATIONS:
Overall Officials: XinYan Bi, PhD, Principal Investigator — Senior Scientist II
Locations (1):
- Clinical Nutrition Research Centre (CNRC), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Access to and the key/password linking participant identifiable data to research data will be handed to a trusted third party (SIFBI HBRO) who is not part of the study team upon the end of data collection. All collected hardcopy data will be filed and stored in secure key-access drawers or in a key access room which will remain locked at all times. These keys are held by SIFBI HBRO and authorized staff at the centre and only study team members and authorized staff are allowed to draw the files. For electronic data, they will be stored in a secured computer that is password protected.

REFERENCES:
- [Background] Ho LH, Bhat R. Exploring the potential nutraceutical values of durian (Durio zibethinus L.) - an exotic tropical fruit. Food Chem. 2015 Feb 1;168:80-9. doi: 10.1016/j.foodchem.2014.07.020. Epub 2014 Jul 11. PMID 25172686
- [Background] Terada Y, Hosono T, Seki T, Ariga T, Ito S, Narukawa M, Watanabe T. Sulphur-containing compounds of durian activate the thermogenesis-inducing receptors TRPA1 and TRPV1. Food Chem. 2014 Aug 15;157:213-20. doi: 10.1016/j.foodchem.2014.02.031. Epub 2014 Feb 15. PMID 24679773
- [Background] Zubairi, S.I., et al., Durian Locule (Endocarp) Water Immersion Drinking Effect to Reduce Heaty Sensation after Flesh Consumption: A Preliminary Study. Current Research in Nutrition and Food Science Journal, 2021. 9(3): p. 866-874.